CLINICAL TRIAL: NCT04690465
Title: Effectiveness of Resistance Training on Resilience in Hong Kong Chinese Older Adults: Study Protocol for a Randomized Controlled Trial
Brief Title: Resistance Training on Elderly Resilience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Sun Yat-sen University (Other); Nanjing Normal University (Other)
Responsible Party: Principal Investigator, Chung Pak Kwong, Professor; Associate Dean (Development) of the Faculty of Social Sciences, Hong Kong Baptist University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: GRF Ref: 12610119
Record Dates: First submitted 2020-12-23; First posted 2020-12-30 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Age Problem; Healthy Aging; Activity, Motor
Keywords: Resistance Training; Older Adults; Ageing; Resilience; Psychological Health
MeSH Terms: conditions — Motor Activity; Psychological Well-Being | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Qualified participants who have signed a consent letter will be randomly assigned into three groups by a draw of lots, in a ratio of 1:1:1. The three groups will be 1) Intervention group: Resistance training (n = 40); 2) Active concurrent control group: Eight-form Yang-style Tai Chi program (n = 40); and 3) Non-treatment control group (n = 40).
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resistance training (Experimental): In the 16 week resistance training, there will be 3 sessions per week, the duration of each session will be 60 minutes, which include 10min of warm-up, 40min of main exercise, and 10min of cool-down. The intensity will be light to somewhat hard (Rating of Perceived Exertion (RPE) 11 to 13; using the Cantonese version of RPE). In resistance training, the weights (resistance) will be from participants' own bodies, dumbbells, and adjustable ankle weights.
  Interventions: Behavioral: Resistance training
- Eight-form Yang-style Tai Chi program (Active Comparator): In Tai Chi, the 16-week program will be divided into cognitive, associated, and automatic stages. The coach will apply a group teaching with individual instruction on specific movements based on participant's needs in skills learning and acquisition. The same training principles of individuality and progression as well as training log-book used in resistance training will also be applied to Tai Chi training program.
  Interventions: Behavioral: Eight-form Yang-style Tai Chi program
- Non-treatment Concurrent Control (No Intervention): Participants in this group will not participate in any specific intervention during the whole study (the 16-week intervention and 12-week follow-up periods), but they will be asked to keep a daily log on their physical activity, medicine used, illness, diet, sleep quality and other health and physical activity related information (e.g., attending healthy eating workshops).

INTERVENTIONS:
Behavioral: Resistance training — Participants will receive a 16-week resistance training program, with 3 times a week (a total of 48 training sessions) and 60 minutes per session intervention, which is adopted from the 12-week resistance training program introduced in the book "Growing Stronger: Strength Training for Older Adults" (Seguin et al., 2002), with minor modifications under the advice of Physical Fitness Association of Hong Kong, China (PFA).
  Other Names: Strength training group
  Arms: Resistance training
Behavioral: Eight-form Yang-style Tai Chi program — The active concurrent control group will receive Eight-form Yang-style Tai Chi program which has been confirmed feasible and will be taught by the qualified coach.
  Other Names: Tai Chi Group
  Arms: Eight-form Yang-style Tai Chi program

SUMMARY:
Background: There is on one hand sufficient evidence showing strong association between resilience and self-rated successful aging. On the other hand, strength training could contribute the cultivation of resilience among older adults. Therefore, the current study aims to examine the effectiveness of resistance training on resilience among Chinese older adults in Hong Kong.

Methods: This study will apply a three-group, double blinded (outcome assessors and data analysts), randomized controlled trial (RCT) to examine the effectiveness of the interventions on resilience, functional fitness, and health related quality of life immediately after a 16-week intervention, as well as the residual effects 12 weeks after completion of the interventions.

Discussion: It is expected that resistance training is promising or even superior to aerobic training in the improvement of resilience. Given the limited evidence on the literature, it is urgently needed to explore the effects of resistance training on the improvement of resilience in older adults. Findings of the current study can contribute to the development of effective resistant training programs for the promotion of resilience among older adults.

ELIGIBILITY:
Inclusion Criteria:

* 65 to 74 years old;
* capable to walk without assistive device;
* apparently healthy and live independently in communities

Exclusion Criteria:

* with cardiovascular or related diseases that prevent from resistance training;
* fail the PAR-Q screening or without physician's advice on readiness of participation in resistance training;
* with substantial experience in practicing resistance training or Tai Chi;
* with high level of resilience.

Ages: 65 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Resilience - The Chinese Version of Resilience Scale | The measure is conducted to examine the change from baseline resilience level at 4 months and at 7 months.
  Chinese version of RS (CRS) will be used to measure participants' resilience in the study. The CRS was modified from the Resilience Scale developed by Wagnild and Young with subsequent validation in Chinese older population and confirmed its four-factor structure: equanimity, meaningfulness, ceaseless self-improvement, and self-reliance. It is a 7-point Likert scale from 1 (highly disagree) to 7 (highly agree), with a greater score mirroring higher level of resilience. Three levels are set, with scores of 145 and above indicating moderate to high resilience, scores from 126 to 144 indicating low to moderate levels of resilience, and scores less than 126 indicating low resilience.

SECONDARY OUTCOMES:
Functional fitness - Senior Fitness Test (SFT): Body Composition | The measure is conducted to examine the change from baseline body composition at 4 months and at 7 months.
  The functional fitness (FF) of participants will be measured using the Senior Fitness Test (SFT) battery. The SFT is a widely used measurement for functional fitness of older adults in the ageing and physical activity area. Within the SFT, the body mass index (BMI) will be used to examine the body composition of the participants.
Functional fitness - Senior Fitness Test (SFT): Muscle Strength | The measure is conducted to examine the change from baseline Muscle Strength and Endurance level at 4 months and at 7 months.
  The functional fitness (FF) of participants will be measured using the Senior Fitness Test (SFT) battery. The SFT is a widely used measurement for functional fitness of older adults in the ageing and physical activity area. Within the SFT, the 30s chair stand test and 30s arm curl test will be used to examine the muscle strength of the participants.
Functional fitness - Senior Fitness Test (SFT): Aerobic Endurance | The measure is conducted to examine the change from baseline aerobic endurance level at 4 months and at 7 months.
  The functional fitness (FF) of participants will be measured using the Senior Fitness Test (SFT) battery. The SFT is a widely used measurement for functional fitness of older adults in the ageing and physical activity area. Within the SFT, 2min step test will be used to examine the aerobic endurance of the participants.
Functional fitness - Senior Fitness Test (SFT): Flexibility | The measure is conducted to examine the change from baseline flexibility at 4 months and at 7 months.
  The functional fitness (FF) of participants will be measured using the Senior Fitness Test (SFT) battery. The SFT is a widely used measurement for functional fitness of older adults in the ageing and physical activity area. Within the SFT, chair sit-and-reach test and back scratch test will be used to examine the flexibility of the participants.
Functional fitness - Senior Fitness Test (SFT): Motor Ability and Balance | The measure is conducted to examine the change from baseline motor ability and balance at 4 months and at 7 months.
  The functional fitness (FF) of participants will be measured using the Senior Fitness Test (SFT) battery. The SFT is a widely used measurement for functional fitness of older adults in the ageing and physical activity area. Within the SFT, 8ft up-and-go test will be used to examine the motor ability and balance of the participants.
Health related quality of life - The Chinese Version of Short Form-36 (C-SF-36) | The measure is conducted to examine the change from baseline quality of life level at 4 months and at 7 months.
  The SF-36 consists of 36 items covering two dimensions-physical health (physical functioning, role limitations due to physical problems, role limitations due to emotional problems, and social functioning) and mental health (mental health, vitality, body pain, and general health perception).

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Baptist University Sports Hall, Hong Kong, Kowloon, Hong Kong

REFERENCES:
- [Derived] Chung PK, Zhang CQ, Zhao Y, Wong MYC, Hu C. Effectiveness of resistance training on resilience in Hong Kong Chinese older adults: study protocol for a randomized controlled trial. BMC Geriatr. 2021 Apr 15;21(1):250. doi: 10.1186/s12877-021-02197-8. PMID 33858336